CLINICAL TRIAL: NCT04459624
Title: Comparison of the Effects of Quadratus Lumborum Block (QLB) and Erector Spina Plane Block (ESP) on Postoperative Pain in Open Nephrectomy
Brief Title: Comparison of Quadratus Lumborum Block and Erector Spina Plane Block in Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Meryem Onay, Specialist Doctor-Anesthesiologist, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ESOGU 2
Record Dates: First submitted 2020-06-23; First posted 2020-07-07 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Pain, Postoperative; Postoperative Complications
Keywords: Erector Spina Plan Block; Quadratus Lumborum Block; Nephrectomy; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Group E: ESP block will be applied at the end of the operation. Patients will receive paracetamol 1gr 4 * 1 and tramadol 1mg/kg 30 minutes before the end of the operation. All patients will undergo IV morphine patient-controlled analgesia (PCA). Pain, opioid consumption, hemodynamic parameters and complications will be monitored in the first 24 hours in the postoperative period.
  Group Q: QLB2 block will be applied at the end of the operation. Patients will receive paracetamol 1gr 4 * 1 and tramadol 1mg / kg 30 minutes before the end of the operation. All patients will undergo IV morphine patient-controlled analgesia (PCA). Pain, opioid consumption, hemodynamic parameters and complications will be monitored in the first 24 hours in the postoperative period.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In the postoperative period, the effectiveness and safety of the block will be evaluated by another researcher (blind) who does not know which group the patient is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP block (Active Comparator): Intervention: Erector Spina Plane Block will administer with 20 ml of % 0.25 bupivacaine
  Interventions: Procedure: Erector Spina Plane Block
- QLB 2 block (Active Comparator): Intervention: Quadratus Lumborum Block 2 will administer with 20 ml of % 0.25 bupivacaine
  Interventions: Procedure: Quadratus Lumborum Block 2

INTERVENTIONS:
Procedure: Erector Spina Plane Block — Group E (ESP block) will be applied 20 ml of % 0.25 bupivacaine between the erector spina muscle and transverse process at the 8th thoracic level. The blocks will be administered under general anesthesia in lateral position by the same anesthesiologist.
  Other Names: Fascial plane block at nephrectomy
  Arms: ESP block
Procedure: Quadratus Lumborum Block 2 — Group Q (QLB2 block) lumbar interfacial triangle (LIFT) will be applied 20 ml of % 0.25 bupivacaine. The blocks will be administered under general anesthesia in lateral position by the same anesthesiologist.
  Other Names: Fascial plane block at nephrectomy
  Arms: QLB 2 block

SUMMARY:
Postoperative pain is important due to the limitation of physical functions, delay in recovery of quality of life, long-term opiate use, length of hospital stay, increased care costs and early postoperative pain trigger chronic pain. It is associated with postoperative morbidity. Multimodal analgesia techniques with fascial plan blocks are frequently used.The investigators aimed to evaluate the effect of QLB2 and ESP on postoperative pain scores in nephrectomy surgery, total opiate consumption, initial analgesia requirement, additional analgesia consumption, patient and surgeon satisfaction.

DETAILED DESCRIPTION:
At the end of the operation, patients will be randomly divided into 2 groups as Group E (ESP block) and Group Q (QLB). The blocks will be administered under general anesthesia in lateral position by same anesthesiologist. Group E (ESP block) will be applied 20 ml of %0.25 bupivacaine between the erector spina muscle and transverse process at the 8th thoracic level. Group Q (QLB2 block) will be applied 20 ml of %0.25 bupivacaine at lumbar interfacial triangle (LIFT). At the end of the operation, the patients with a Modified aldreate score ≥9 will be sent from the postoperative anesthesia unit. All patients will be equipped with an IV morphine patient-controlled analgesia (PCA) device. The solution will be prepared such that morphine is 0.5 mg / ml. PCA 1mg bolus dose will be delivered with 10 min lock-out time. In the postoperative period, the patient was evaluated by another researcher who blind to the groups at the 1st and 6th, 12th and 24th hours. Visual pain scores (VAS) in rest and movement, hemodynamic values, morphine consumption, initial analgesic requirement, nausea-vomiting score, ramsey sedation scale, length of hospital stay, patient and surgeon satisfaction, and postoperative complications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Partial or radical nephrectomy
* American Society of Anesthesiologist physical status I-III

Exclusion Criteria:

* Infection in the incision area
* Coagulation disorder
* Known allergy history against to the study drugs
* Lack of adequate cognitive activity in the use of patient-controlled analgesia and VAS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Effect of QLB2 and ESP on postoperative pain scores in nephrectomy surgery | 24 hours
  Visual analog scale at rest and movement (0 (no pain)-10 (unbearable pain))

SECONDARY OUTCOMES:
Total opiate consumption | 24 hours
  Total morphine patient control analgesia prepared 0.5 mg / ml. PCA 1mg bolus dose will be delivered with 10 min lock-out time. Follow up morphine consumption at postoperative 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Onay, Dr, Principal Investigator — Eskisehir Osmangazi University Faculty Of Medicine
Locations (1):
- Eskisehir Osmangazi Univercıty, Odunpazari, Eskişehir, Turkey (Türkiye)

REFERENCES:
- [Background] Aksu C, Sen MC, Akay MA, Baydemir C, Gurkan Y. Erector Spinae Plane Block vs Quadratus Lumborum Block for pediatric lower abdominal surgery: A double blinded, prospective, and randomized trial. J Clin Anesth. 2019 Nov;57:24-28. doi: 10.1016/j.jclinane.2019.03.006. Epub 2019 Mar 6. PMID 30851499
- [Background] Ueshima H, Otake H, Lin JA. Ultrasound-Guided Quadratus Lumborum Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:2752876. doi: 10.1155/2017/2752876. Epub 2017 Jan 3. PMID 28154824
- [Background] Oksuz G, Bilal B, Gurkan Y, Urfalioglu A, Arslan M, Gisi G, Oksuz H. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block in Children Undergoing Low Abdominal Surgery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2017 Sep/Oct;42(5):674-679. doi: 10.1097/AAP.0000000000000645. PMID 28759502
- [Background] Yousef NK. Quadratus Lumborum Block versus Transversus Abdominis Plane Block in Patients Undergoing Total Abdominal Hysterectomy: A Randomized Prospective Controlled Trial. Anesth Essays Res. 2018 Jul-Sep;12(3):742-747. doi: 10.4103/aer.AER_108_18. PMID 30283187